CLINICAL TRIAL: NCT00218829
Title: Dimethylsulphoxide-supported Photodynamic Therapy of Basal Cell Carcinoma Combined With Curettage - A 6 Year Clinical and Histological Evaluation.
Brief Title: DMSO-PDT of BCC - A 6 Year Follow up
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: EC-002
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Basal Cell
Keywords: Photodynamic treatment; Basal cell carcinoma; DMSO
MeSH Terms: conditions — Carcinoma, Basal Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to registrate long time clinical and histological treatment response of basal cell carcinoma (BCC) lesions treated with one or two procedures of dimethylsulfoxide supported 5-aminolaevulinic acid photodynamic therapy (DMSO-PDT).

ELIGIBILITY:
Inclusion Criteria:

* histological verified bcc.
* one or two PDT treatments with treatment interval no longer than two weeks.
* lesion complete response three months after therapy.

Exclusion Criteria:

* pregnant.
* Gorlin's syndrome.
* morpheaform or pigmented bcc.
* histology older than one year.
* tumour infiltration more than four mm.
* previous PDT treated lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 1997-09 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eidi Christensen, MD, Principal Investigator — St. Olav University Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Christensen E, Skogvoll E, Viset T, Warloe T, Sundstrom S. Photodynamic therapy with 5-aminolaevulinic acid, dimethylsulfoxide and curettage in basal cell carcinoma: a 6-year clinical and histological follow-up. J Eur Acad Dermatol Venereol. 2009 Jan;23(1):58-66. doi: 10.1111/j.1468-3083.2008.02946.x. Epub 2008 Sep 18. PMID 18803580